CLINICAL TRIAL: NCT02268253
Title: Tagraxofusp (SL-401) in Patients With Chronic Myelomonocytic Leukemia (CMML)
Brief Title: Tagraxofusp (SL-401) in Participants With Chronic Myelomonocytic Leukemia (CMML) and Myelofibrosis (MF)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stemline Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STML-401-0314
Record Dates: First submitted 2014-10-10; First posted 2014-10-20 (Estimated); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Myelofibrosis; Chronic Myelomonocytic Leukemia
Keywords: MF; CMML; CMML-1; CMML-2
MeSH Terms: conditions — Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic | interventions — tagraxofusp

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Dose Level 1 - Tagraxofusp - 7 micrograms/kilogram (µg/kg)/day - Chronic Myelomonocytic Leukemia (Experimental)
  Interventions: Drug: Tagraxofusp Injection
- Dose Level 2 - Tagraxofusp - 9 µg/kg/day - Chronic Myelomonocytic Leukemia (Experimental)
  Interventions: Drug: Tagraxofusp Injection
- Dose Level 3 - Tagraxofusp - 12 µg/kg/day - Chronic Myelomonocytic Leukemia (Experimental)
  Interventions: Drug: Tagraxofusp Injection
- Dose Level 1 - Tagraxofusp - 7 µg/kg/day - Myelofibrosis (Experimental)
  Interventions: Drug: Tagraxofusp Injection
- Dose Level 2 - Tagraxofusp - 9 µg/kg/day - Myelofibrosis (Experimental)
  Interventions: Drug: Tagraxofusp Injection
- Dose Level 3 - Tagraxofusp - 12 µg/kg/day - Myelofibrosis (Experimental)
  Interventions: Drug: Tagraxofusp Injection

INTERVENTIONS:
Drug: Tagraxofusp Injection — Tagraxofusp was administered as a 15-minute intravenous infusion once daily for the first 3 consecutive days of each dosing cycle.
  Other Names: SL-401; Elzonris

SUMMARY:
This multicenter, multi-arm trial evaluated the safety and efficacy of tagraxofusp, a cell division cycle protein 123 homolog-targeted therapy, in participants with either CMML or MF. There were 2 CMML cohorts, 1 enrolled participant with CMML (CMML-1 or CMML-2) who were refractory/resistant or intolerant to hypomethylating agents (HMA), hydroxyurea (HU), or intensive chemotherapy and 1 enrolled treatment-naive participants with CMML (CMML-1 or CMML-2) with molecular features associated with poor prognosis. The MF cohort enrolled participants who were resistant/refractory or intolerant to approved Janus kinase (JAK) therapy (JAK1/JAK2 or JAK2).

DETAILED DESCRIPTION:
This was a non-randomized, open-label, multicenter study, divided into 3 stages.

Stage 1: Stage 1 of the study was to enroll participants with CMML, MF, advanced systemic mastocytosis, or advanced symptomatic primary eosinophilic disorder.

Stage 2: Stage 2 was to enroll MF and CMML participants.

Stage 3A: Stage 3A was to enroll 2 populations of participants with CMML, those with CMML-1 or CMML-2 who were refractory/resistant/intolerant to HMAs, HU, or intensive chemotherapy (relapsed/refractory participants); and participants with treatment-naïve CMML-1 or CMML-2 (previously untreated participants) with molecular features associated with a poor prognosis.

ELIGIBILITY:
Key Inclusion Criteria:

All Participants - Participants meeting all the following criteria were considered for enrollment:

1. The participant had a life expectancy of > 6 months.
2. The participant had an Eastern Cooperative Oncology Group performance status of 0-2.
3. The participant had adequate baseline organ function, including cardiac, renal, and hepatic function:

   * Left ventricular ejection fraction 2: institutional lower limit of normal as measured by multigated acquisition scan or 2-dimensional echocardiogram within 28 days prior to the start of therapy and no clinically significant abnormalities on a 12-lead electrocardiogram.
   * Serum creatinine ≤ 1.5 milligrams/deciliter (dL).
   * Serum albumin ≥ 3.2 grams (g)/dL (or 32 g/liter [L]) in the absence of receipt of intravenous albumin within the previous 72 hours.
   * Aspartate transaminase and alanine transaminase ≤ 2.5 times the upper limit of normal (ULN).
   * Creatine phosphokinase ≤ 2.5 times the ULN.
   * Absolute neutrophil count ≥ 0.5×10^9/L.
4. If a woman of child-bearing potential, the participant had a negative serum or urine pregnancy test within 1 week prior to tagraxofusp treatment (intervals shorter than 1 week are acceptable, if required by institutional guidelines).
5. The participant (either male or female) agrees to use acceptable contraceptive methods for the duration of time in the study, and to continue to use acceptable contraceptive methods for 1 week after the last tagraxofusp infusion.
6. The participant can adhere to the study visit schedule and other protocol requirements, including follow-up for response assessments.

Myelofibrosis (Stage 2) - Participants with MF meeting all of the following criteria, in addition to those specified for all participants, above, are eligible for enrollment in Stage 2:

1. Participant meets the 2016 World Health Organization (WHO) diagnostic criteria for MF and has an International Prognostic Scoring System/Dynamic International Prognostic Scoring System (IPSS/DIPSS)/DIPSS-plus intermediate-2 or high-risk disease. Participants with IPSS/DIPSS/DIPSS-plus low or intermediate-1 risk disease who have at least 1 of the following symptoms are also eligible: MF-related anemia (hemoglobin < 10 g/dL), splenomegaly (palpable size > 10 centimeters), leukocytosis (white blood cell count [WBC] > 25×10^9/L), marked thrombocytosis (platelet count > 1,000×10^9/L), or constitutional symptoms (weight loss > 10%, during prior 6 months or fever [> 37.5 degrees Celsius or drenching night sweats for > 6 weeks]), as recommended by the European LeukemiaNet/International Working Group (ELN/IWG) 2018 criteria.
2. Participant was approved JAK therapy (JAK1/JAK2 or JAK2) resistant/refractory or intolerant, in accordance with the ELN/IWG 2018 criteria, and at least 4 weeks have elapsed between the last dose of any MF-directed drug treatments, excluding HU, and study enrollment (first dose). HU can be continued until 2 weeks prior to study enrollment.
3. Participant was not eligible for an immediate allogeneic-stem cell transplantation.

   CMML (Stage 3A):
4. Participant had a 2016 WHO-defined diagnosis of CMML (persistent monocytosis ≥ 1×10^9/L for at least 3 months, with other causes excluded, and monocytes ≥10% of WBC in peripheral blood, no criteria and no previous history of CMML, essential thrombocythemia, polycythemia vera, and acute promyelocytic leukemia; if eosinophilic, neither platelet-derived growth factor receptor A, platelet-derived growth factor receptor beta, fibroblast growth factor receptor 1 rearrangements nor pericentriolar material 1-JAK2 translocation; < 20% blasts in peripheral blood and bone marrow aspirate; > 1 following criteria: dysplasia in > 1 myeloid lineage, acquired clonal cytogenetic or molecular abnormality in hematopoietic cells).
5. Participant had 2016 WHO-defined CMML-1 (2-4% blasts in peripheral blood and/or 5-9% blasts in bone marrow) and CMML-2 (5-19% blasts in peripheral blood and/or 10-19% blasts in bone marrow, and/or presence of Auer rods).
6. Participant was refractory/resistant/intolerant, as defined for the purposes of this study (in the absence of a standard definition for CMML) below, to HMAs, HU, or intensive chemotherapy, including:

   * Resistance/intolerance to HU is defined as:

     * Uncontrolled myeloproliferation, (platelets > 400×10^9/L and WBC > 10×10^9/L after 3 months of at least 2 g/day of HU); or
     * Myelosuppression at a clinically relevant dose; or
     * Presence of unacceptable HU-related non-hematological toxicities, such as mucocutaneous manifestations, gastrointestinal symptoms, pneumonitis, or fever at any dose of HU.
   * Conventional definition for HMA failure is defined for the purposes of this study (in the absence of a standard definition for CMML) as:

     * Disease progression following at least 4 to 6 cycles of 5-azacitidine or decitabine; or
     * Relapse after achieving response; or
     * Intolerance to 5-azacitidine or decitabine at the prescribed dose.

   or

   • Participant was classified as high-risk based on the presence of morphological features, as described by the 2016 WHO prognostic system, and the clinical and molecular features described in molecularly integrated prognostic systems, such as the Groupe Français des Myélodysplasies, Mayo Molecular Model, and the CMML specific prognostic model and thus is not expected to benefit from HMAs.
7. Participant was ineligible for an immediate allogeneic stem cell transplantation (allo-SCT).

Key Exclusion Criteria:

1. Participant had persistent clinically significant toxicities Grade ≥2 from previous therapies, including cytotoxic chemotherapy, targeted therapies, biological therapies, or immunotherapies, not readily controlled by supportive measures (excluding alopecia, nausea, and fatigue).
2. Participant received treatment with any disease-related therapy, including radiation therapy within 14 days of study entry.
3. Participant received an allo-SCT within 3 months of study entry.
4. Participant received treatment with another investigational agent within 14 days of study entry or concurrent treatment with another investigational agent.
5. Participant previously received treatment with tagraxofusp or has a known hypersensitivity to any components of the drug product.
6. Participant had an active malignancy and/or cancer history (excluding myeloproliferative disorders and concomitant myeloid malignancies as specified in the inclusion criteria) that could confound the assessment of the study endpoints.
7. Participant had clinically significant cardiovascular disease (for example, uncontrolled or any New York Heart Association Class 3 or 4 congestive heart failure, uncontrolled angina, history of myocardial infarction, unstable angina, or stroke within 6 months prior to study entry, uncontrolled hypertension or clinically significant arrhythmias not controlled by medication).
8. Participant had uncontrolled, clinically significant pulmonary disease (for example, chronic obstructive pulmonary disease, pulmonary hypertension) that, in the Investigator's opinion, would have put the participant at significant risk for pulmonary complications during the study.
9. Participant had known active or suspected disease involvement of the central nervous system (CNS). If suspected due to clinical findings, CNS disease was to be ruled out with relevant imaging and/or examination of cerebrospinal fluid.

Note: Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (22):
  - University of California, San Francisco, Clovis, California
  - City of Hope, Duarte, California
  - University of California, Los Angeles, Los Angeles, California
  - Stanford Cancer Institute, Stanford, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Indiana Blood and Bone Marrow Transplantation, Indianapolis, Indiana
  - University of Kansas Cancer Center, Westwood, Kansas
  - Norton Cancer Institute, Louisville, Kentucky
  - Dana Farber Cancer Institute (DFCI), Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - John Theurer Cancer Center, Hackensack, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medical Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario

REFERENCES:
- [Derived] Yacoub A, Ali H, Gupta V, Wang ES, Patnaik MM, Schiller GJ, Taparia M, Mughal TI, Lindsay R, Galleu A, Gupta I, Pemmaraju N. Final safety and efficacy results from a phase 1/2 study of tagraxofusp, a CD123-targeted therapy, for myelofibrosis. Blood Neoplasia. 2025 Aug 25;2(4):100165. doi: 10.1016/j.bneo.2025.100165. eCollection 2025 Nov. PMID 41146971
- [Derived] Patnaik MM, Ali H, Wang ES, Yacoub A, Foran JM, Gupta V, Schiller GJ, Stevens DA, Talpaz M, Wall S, Lasho TL, Mangaonkar AA, Badar T, Lindsay R, Galleu A, Gupta I, Pemmaraju N, Garcia-Manero G. Tagraxofusp, a CD123-targeted therapy, for chronic myelomonocytic leukemia: final results of a phase 1/2 study. Blood Neoplasia. 2025 May 11;2(4):100115. doi: 10.1016/j.bneo.2025.100115. eCollection 2025 Nov. PMID 40919483

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1 - Tagraxofusp - 7 Micrograms/Kilogram (µg/kg)/Day - Chronic Myelomonocytic Leukemia: Tagraxofusp was administered as a 15-minute intravenous (IV) infusion once daily for the first 3 consecutive days of each dosing cycle.
- Dose Level 2 - Tagraxofusp - 9 µg/kg/Day - Chronic Myelomonocytic Leukemia; Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Chronic Myelomonocytic Leukemia; Dose Level 1 - Tagraxofusp - 7 µg/kg/Day - Myelofibrosis; Dose Level 2 - Tagraxofusp - 9 µg/kg/Day - Myelofibrosis; Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Myelofibrosis; Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Advanced Systemic Mastocytosis: Tagraxofusp was administered as a 15-minute IV infusion once daily for the first 3 consecutive days of each dosing cycle.
Period: Stage 1
Arm/Group | Dose Level 1 - Tagraxofusp - 7 Micrograms/Kilogram (µg/kg)/Day - Chronic Myelomonocytic Leukemia | Dose Level 2 - Tagraxofusp - 9 µg/kg/Day - Chronic Myelomonocytic Leukemia | Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Chronic Myelomonocytic Leukemia | Dose Level 1 - Tagraxofusp - 7 µg/kg/Day - Myelofibrosis | Dose Level 2 - Tagraxofusp - 9 µg/kg/Day - Myelofibrosis | Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Myelofibrosis | Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Advanced Systemic Mastocytosis
Started | 1 | 2 | 2 | 2 | 1 | 1 | 0
Received At Least 1 Dose of Study Drug (Safety Population) | 1 | 2 | 2 | 2 | 1 | 1 | 0
Treatment Naïve (Modified Intent-to-Treat) (Received at least 1 dose of study drug and was evaluable for efficacy assessment) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Relapsed/Refractory (Modified Intent-to-Treat) (Received at least 1 dose of study drug and was evaluable for efficacy assessment) | 0 | 1 | 2 | 2 | 0 | 1 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 2 | 2 | 2 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 2 | 2 | 2 | 1 | 1 | 0
Period: Stage 2
Arm/Group | Dose Level 1 - Tagraxofusp - 7 Micrograms/Kilogram (µg/kg)/Day - Chronic Myelomonocytic Leukemia | Dose Level 2 - Tagraxofusp - 9 µg/kg/Day - Chronic Myelomonocytic Leukemia | Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Chronic Myelomonocytic Leukemia | Dose Level 1 - Tagraxofusp - 7 µg/kg/Day - Myelofibrosis | Dose Level 2 - Tagraxofusp - 9 µg/kg/Day - Myelofibrosis | Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Myelofibrosis | Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Advanced Systemic Mastocytosis
Started | 0 | 0 | 24 (Participants enrolled into Stage 2 only. Participants from Stage 1 did not roll over into Stage 2.) | 0 | 0 | 35 (Participants enrolled into Stage 2 only. Participants from Stage 1 did not roll over into Stage 2.) | 1 (Participant enrolled into Stage 2 only.)
Received At Least 1 Dose of Study Drug (Safety Population) | 0 | 0 | 24 | 0 | 0 | 35 | 1
Treatment Naïve (Modified Intent-to-Treat) (Received at least 1 dose of study drug and was evaluable for efficacy assessment) | 0 | 0 | 8 | 0 | 0 | 5 | 0
Relapsed/Refractory (Modified Intent-to-Treat) (Received at least 1 dose of study drug and was evaluable for efficacy assessment) | 0 | 0 | 15 | 0 | 0 | 24 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 24 | 0 | 0 | 35 | 1
Not completed — Disease Recurrence/ Progression | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 0 | 2 | 0
Not completed — Completion of 7 or More Cycles of Treatment | 0 | 0 | 2 | 0 | 0 | 7 | 0
Not completed — Death | 0 | 0 | 19 | 0 | 0 | 20 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 4 | 0
Not completed — Transferred to Hospice | 0 | 0 | 0 | 0 | 0 | 2 | 0
Period: Stage 3A
Arm/Group | Dose Level 1 - Tagraxofusp - 7 Micrograms/Kilogram (µg/kg)/Day - Chronic Myelomonocytic Leukemia | Dose Level 2 - Tagraxofusp - 9 µg/kg/Day - Chronic Myelomonocytic Leukemia | Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Chronic Myelomonocytic Leukemia | Dose Level 1 - Tagraxofusp - 7 µg/kg/Day - Myelofibrosis | Dose Level 2 - Tagraxofusp - 9 µg/kg/Day - Myelofibrosis | Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Myelofibrosis | Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Advanced Systemic Mastocytosis
Started | 0 | 0 | 13 (Participants enrolled into Stage 3A only. Participants from Stage 2 did not roll over into Stage 3A.) | 0 | 0 | 0 | 0
Received At Least 1 Dose of Study Drug (Safety Population) | 0 | 0 | 13 | 0 | 0 | 0 | 0
Treatment Naïve (Modified Intent-to-Treat) (Received at least 1 dose of study drug and was evaluable for efficacy assessment) | 0 | 0 | 7 | 0 | 0 | 0 | 0
Relapsed/Refractory (Modified Intent-to-Treat) (Received at least 1 dose of study drug and was evaluable for efficacy assessment) | 0 | 0 | 5 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 13 | 0 | 0 | 0 | 0
Not completed — Disease Recurrence/ Progression | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 5 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who received at least 1 dose of study drug.
Groups:
- Dose Level 1 -Tagraxofusp - 7 µg/kg/Day - Chronic Myelomonocytic Leukemia; Dose Level 2 - Tagraxofusp - 9 µg/kg/Day - Chronic Myelomonocytic Leukemia; Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Chronic Myelomonocytic Leukemia; Dose Level 1 - Tagraxofusp - 7 µg/kg/Day - Myelofibrosis; Dose Level 2 - Tagraxofusp - 9 µg/kg/Day - Myelofibrosis; Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Myelofibrosis; Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Advanced Systemic Mastocytosis: Tagraxofusp was administered as a 15-minute IV infusion once daily for the first 3 consecutive days of each dosing cycle.
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 -Tagraxofusp - 7 µg/kg/Day - Chronic Myelomonocytic Leukemia | Dose Level 2 - Tagraxofusp - 9 µg/kg/Day - Chronic Myelomonocytic Leukemia | Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Chronic Myelomonocytic Leukemia | Dose Level 1 - Tagraxofusp - 7 µg/kg/Day - Myelofibrosis | Dose Level 2 - Tagraxofusp - 9 µg/kg/Day - Myelofibrosis | Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Myelofibrosis | Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Advanced Systemic Mastocytosis | Total
Number analyzed (Participants) | 1 | 2 | 39 | 2 | 1 | 36 | 1 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (NA) — Insufficient number of participants to determine standard deviation. | 66.0 (4.24) | 69.1 (8.88) | 65.5 (4.95) | 81.0 (NA) — Insufficient number of participants to determine standard deviation. | 70.4 (7.97) | 63 (NA) — Insufficient number of participants to determine standard deviation. | 69.3 (8.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 10 | 1 | 1 | 16 | 0 | 29
  Male | 1 | 1 | 29 | 1 | 0 | 20 | 1 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 4 | 0 | 0 | 5 | 0 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 5
  White | 0 | 1 | 32 | 2 | 1 | 25 | 1 | 62
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 4
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status is a scale that measures how cancer affects a participant's daily living activities. The scale ranges from 0 (normal activity) to 5 (dead). 0 = Fully active without restriction; 1 = Restricted in physically strenuous activity; 2 = Ambulatory, capable of all selfcare; 3 = Capable of limited selfcare; 4 = Completely disabled; 5 = Dead.
  Participants
    0 | 0 | 0 | 5 | 1 | 0 | 3 | 0 | 9
    1 | 1 | 2 | 29 | 0 | 1 | 23 | 1 | 57
    2 | 0 | 0 | 5 | 1 | 0 | 10 | 0 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: During Stage 1, DLT was defined as any of the following occurring during the first cycle of therapy: any treatment-emergent Grade 4 transaminase or creatine phosphokinase (CPK) elevation (confirmed within 24 hours of initial identification), regardless of duration or relationship to SL-401; any Grade ≥3 non-hematologic toxicity (unrelated to underlying MPN), with the exception of Grade 3 laboratory toxicities that resolve to Grade ≤1 or baseline ≤28 days after the last infusion of SL-401, or the following Grade 3 toxicities if they resolve to Grade ≤1 or baseline ≤21 days after the last infusion of SL-401, arthralgia, myalgia, fever responding to treatment, nausea and/or vomiting (excluding cases that require tube feeding, total parenteral nutrition, or hospitalization) or diarrhea associated with suboptimal prophylaxis or treatment; Grade 4 neutropenia or Grade 4 thrombocytopenia with a duration (at Grade 4) of ≥28 days.
Time Frame: 21 days of Cycle 1 (21 days/cycle)
Population: Safety Population: All participants who received at least 1 dose of study drug during Stage 1 only. 'Dose Level 3 - Tagraxofusp - 12 μg/kg/Day - Advanced Systemic Mastocytosis' arm enrolled during Stage 2. Here, 'Overall Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure in Stage 1 only.
Measure: Number; unit: participants
Groups:
- Dose Level 1 - Tagraxofusp - 7 µg/kg/Day - Chronic Myelomonocytic Leukemia; Dose Level 2 - Tagraxofusp - 9 µg/kg/Day - Chronic Myelomonocytic Leukemia; Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Chronic Myelomonocytic Leukemia; Dose Level 1 - Tagraxofusp - 7 µg/kg/Day - Myelofibrosis; Dose Level 2 - Tagraxofusp - 9 µg/kg/Day - Myelofibrosis; Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Myelofibrosis: Tagraxofusp was administered as a 15-minute IV infusion once daily for the first 3 consecutive days of each dosing cycle.
Arm/Group | Dose Level 1 - Tagraxofusp - 7 µg/kg/Day - Chronic Myelomonocytic Leukemia | Dose Level 2 - Tagraxofusp - 9 µg/kg/Day - Chronic Myelomonocytic Leukemia | Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Chronic Myelomonocytic Leukemia | Dose Level 1 - Tagraxofusp - 7 µg/kg/Day - Myelofibrosis | Dose Level 2 - Tagraxofusp - 9 µg/kg/Day - Myelofibrosis | Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Myelofibrosis
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 1 | 1
participants | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants (responders) who achieved disease-specific complete response (CR) or partial response (PR) after treatment. For response assessment of myelofibrosis during both Stage 1 and Stage 2, the International Working Group-Myeloproliferative Neoplasms Research and Treatment and European LeukemiaNet (IWG-MRT/ELN 2013) criteria were used. For chronic myelomonocytic leukemia, during both Stage 1 and Stage 2, the International Working Group 2006 response criteria for myelodysplastic syndromes (IWG MDS 2006) were used for response assessment while the Myelodysplastic/Myeloproliferative Neoplasms (MDS/MPN) 2015 criteria were used for response assessment during Stage 3A.
Time Frame: 1145 days
Population: Modified Intent-to-Treat (mITT): Any participant who received at least 1 dose of study intervention and was evaluable for efficacy assessment. Presentation of reporting groups based upon shared criteria used for response assessment and prior treatment history (previously untreated [treatment naive]; previously treated [relapsed/refractory]). Here, 'Overall Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- Stages 1-2: Tagraxofusp 12 µg/kg/Day - Treatment Naive - Myelofibrosis: Treatment-naive participants with myelofibrosis treated with tagraxofusp 12 µg/kg/day.
- Stages 1-2: Tagraxofusp 12 µg/kg/Day - Relapsed/Refractory - Myelofibrosis: Relapsed/refractory participants with myelofibrosis treated with tagraxofusp 12 µg/kg/day.
- Stages 1-2: Tagraxofusp 12 µg/kg/Day - Treatment Naive - Chronic Myelomonocytic Leukemia; Stage 3A: Tagraxofusp 12 µg/kg/Day - Treatment Naive - Chronic Myelomonocytic Leukemia: Treatment-naive participants with chronic myelomonocytic leukemia treated with tagraxofusp 12 µg/kg/day.
- Stages 1-2: Tagraxofusp 12 µg/kg/Day - Relapsed/Refractory - Chronic Myelomonocytic Leukemia; Stage 3A: Tagraxofusp 12 µg/kg/Day - Relapsed/Refractory - Chronic Myelomonocytic: Relapsed/refractory participants with chronic myelomonocytic leukemia treated with tagraxofusp 12 µg/kg/day.
Arm/Group | Stages 1-2: Tagraxofusp 12 µg/kg/Day - Treatment Naive - Myelofibrosis | Stages 1-2: Tagraxofusp 12 µg/kg/Day - Relapsed/Refractory - Myelofibrosis | Stages 1-2: Tagraxofusp 12 µg/kg/Day - Treatment Naive - Chronic Myelomonocytic Leukemia | Stages 1-2: Tagraxofusp 12 µg/kg/Day - Relapsed/Refractory - Chronic Myelomonocytic Leukemia | Stage 3A: Tagraxofusp 12 µg/kg/Day - Treatment Naive - Chronic Myelomonocytic Leukemia | Stage 3A: Tagraxofusp 12 µg/kg/Day - Relapsed/Refractory - Chronic Myelomonocytic
Number analyzed (Participants) | 5 | 25 | 8 | 17 | 7 | 5
participants | 0 [NA to NA] — Not estimable due to no responders | 1 [0.1 to 20.4] | 0 [NA to NA] — Not estimable due to no responders | 0 [NA to NA] — Not estimable due to no responders | 1 [0.4 to 57.9] | 0 [NA to NA] — Not estimable due to no responders

ADVERSE EVENTS:
Time Frame: Up to 1145 days
Description: All reported safety data based upon Safety Population: All participants who received at least 1 dose of study drug.
Arm/Group | Dose Level 1 - Tagraxofusp - 7 µg/kg/Day - Chronic Myelomonocytic Leukemia | Dose Level 2 - Tagraxofusp - 9 µg/kg/Day - Chronic Myelomonocytic Leukemia | Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Chronic Myelomonocytic Leukemia | Dose Level 1 - Tagraxofusp - 7 µg/kg/Day - Myelofibrosis | Dose Level 2 - Tagraxofusp - 9 µg/kg/Day - Myelofibrosis | Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Myelofibrosis | Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Advanced Systemic Mastocytosis
All-Cause Mortality (participants affected / at risk) | 0/1 | 2/2 | 26/39 | 2/2 | 1/1 | 21/36 | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/2 | 23/39 | 1/2 | 1/1 | 20/36 | 1/1
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 39/39 | 2/2 | 1/1 | 35/36 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Dose Level 1 - Tagraxofusp - 7 µg/kg/Day - Chronic Myelomonocytic Leukemia (N=1) | Dose Level 2 - Tagraxofusp - 9 µg/kg/Day - Chronic Myelomonocytic Leukemia (N=2) | Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Chronic Myelomonocytic Leukemia (N=39) | Dose Level 1 - Tagraxofusp - 7 µg/kg/Day - Myelofibrosis (N=2) | Dose Level 2 - Tagraxofusp - 9 µg/kg/Day - Myelofibrosis (N=1) | Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Myelofibrosis (N=36) | Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Advanced Systemic Mastocytosis (N=1)
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 3 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 3 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 6 | 0 | 0 | 3 | 0
Embolism (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Parotitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal cavity packing (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Orchitis (Infections and infestations) | 0 | 0/1 | 0/29 | 0/1 | 0 | 1/20 | 0 — Adverse event only affected male participants.
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulvitis (Infections and infestations) | 0/0 | 0/1 | 0/10 | 0/1 | 0 | 1/16 | 0/0 — Adverse event only affected female participants.
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dementia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laryngeal injury (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematotympanum (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 - Tagraxofusp - 7 µg/kg/Day - Chronic Myelomonocytic Leukemia (N=1) | Dose Level 2 - Tagraxofusp - 9 µg/kg/Day - Chronic Myelomonocytic Leukemia (N=2) | Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Chronic Myelomonocytic Leukemia (N=39) | Dose Level 1 - Tagraxofusp - 7 µg/kg/Day - Myelofibrosis (N=2) | Dose Level 2 - Tagraxofusp - 9 µg/kg/Day - Myelofibrosis (N=1) | Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Myelofibrosis (N=36) | Dose Level 3 - Tagraxofusp - 12 µg/kg/Day - Advanced Systemic Mastocytosis (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 17 | 2 | 1 | 8 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 11 | 1 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 9 | 1 | 0 | 9 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 2 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 6 | 0 | 0 | 3 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 5 | 0 | 0 | 2 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Vision blurred (Eye disorders) | 0 | 0 | 4 | 0 | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 5 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 4 | 0 | 0 | 8 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 14 | 0 | 0 | 10 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 14 | 1 | 0 | 9 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 4 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 5 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 4 | 0 | 0 | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 17 | 1 | 0 | 15 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 3 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 10 | 1 | 0 | 10 | 0
Asthenia (General disorders) | 0 | 0 | 5 | 0 | 0 | 6 | 0
Chest discomfort (General disorders) | 0 | 0 | 4 | 0 | 0 | 3 | 0
Chest pain (General disorders) | 0 | 0 | 4 | 0 | 0 | 5 | 0
Chills (General disorders) | 0 | 0 | 11 | 0 | 0 | 10 | 0
Early satiety (General disorders) | 0 | 0 | 2 | 0 | 0 | 4 | 0
Fatigue (General disorders) | 0 | 1 | 18 | 1 | 0 | 9 | 1
Gait disturbance (General disorders) | 0 | 0 | 4 | 0 | 0 | 2 | 0
Generalised oedema (General disorders) | 0 | 0 | 2 | 0 | 0 | 2 | 0
Influenza like illness (General disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 0
Nodule (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 2 | 1 | 0 | 2 | 0
Oedema (General disorders) | 0 | 0 | 2 | 0 | 0 | 3 | 0
Oedema peripheral (General disorders) | 0 | 2 | 12 | 1 | 1 | 12 | 0
Pain (General disorders) | 0 | 1 | 7 | 0 | 0 | 3 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 0
Pyrexia (General disorders) | 0 | 0 | 10 | 1 | 0 | 11 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 4 | 0 | 0 | 2 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Sepsis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 3 | 0 | 0 | 5 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 4 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 5 | 0 | 0 | 4 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 4 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 2 | 0 | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 11 | 0 | 0 | 8 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 9 | 0 | 0 | 6 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 4 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 2 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 9 | 0 | 0 | 4 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 9 | 0 | 0 | 3 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Weight decreased (Investigations) | 0 | 0 | 3 | 0 | 0 | 5 | 0
Weight increased (Investigations) | 0 | 0 | 12 | 0 | 0 | 8 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 15 | 0 | 0 | 11 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 3 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 0 | 2 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 8 | 0 | 0 | 6 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 5 | 0 | 0 | 2 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 4 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 5 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 18 | 0 | 0 | 17 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 7 | 0 | 0 | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 17 | 0 | 0 | 8 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0 | 0 | 6 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0 | 0 | 3 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 6 | 0 | 0 | 2 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 8 | 1 | 0 | 7 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 14 | 0 | 0 | 4 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 0 | 0 | 3 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 0 | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 0 | 0 | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 8 | 0 | 0 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 0 | 0 | 5 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 9 | 0 | 0 | 11 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 11 | 0 | 0 | 10 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 3 | 1 | 0 | 4 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 4 | 0 | 0 | 6 | 0
Depression (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 2 | 0
Emotional distress (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 9 | 1 | 0 | 6 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 9 | 0 | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 3 | 0 | 0 | 2 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 15 | 1 | 0 | 6 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 12 | 1 | 1 | 13 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 6 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 0 | 0 | 6 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0 | 0 | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 0 | 0 | 2 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 0 | 0 | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 0 | 0 | 5 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 3 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 2 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 3 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 1 | 3 | 0 | 0 | 1 | 1
Embolism (Vascular disorders) | 0 | 0 | 4 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 2 | 1 | 0 | 4 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 0
Hypertension (Vascular disorders) | 0 | 0 | 5 | 0 | 0 | 3 | 1
Hypotension (Vascular disorders) | 0 | 0 | 9 | 0 | 1 | 10 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Petechiae (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hiccups (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
1. Individual site results may be submitted for publication only after the results of the multicenter study are published, 12 months after study completion at all sites, or notification from Stemline that submission of a multicenter publication is no longer planned.
2. Thereafter, the PI is free to publish the results.
3. The PI is required to furnish Stemline with a copy of any proposed publication or presentation for review and comment at least thirty (30) days prior to submission.

DOCUMENTS (2):
  • Study Protocol (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT02268253/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT02268253/SAP_001.pdf